CLINICAL TRIAL: NCT04153955
Title: Earlier Mobilization Post Acute Thrombectomy
Acronym: EMPATHY-II
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never started/initiated.
Sponsor: Brian Silver (Other)
Responsible Party: Sponsor-Investigator, Brian Silver, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00018239
Record Dates: First submitted 2019-10-21; First posted 2019-11-06 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic
Keywords: Mobilization; Thrombectomy; Ischemia; Cerebrovascular Disorders; Brain Diseases; Recovery
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ischemia; Cerebrovascular Disorders; Brain Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors blind to the subject's treatment/arm will do the evaluations at 90 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-Hour Bed Rest (Experimental): Subjects will be mobilized 12 hours after undergoing thrombectomy per usual care
  Interventions: Behavioral: Mobilization
- 24-Hour Bed Rest (Active Comparator): Subjects will be mobilized 24 hours after undergoing thrombectomy per usual care
  Interventions: Behavioral: Mobilization

INTERVENTIONS:
Behavioral: Mobilization — Any movement out of bed

SUMMARY:
This is a phase III trial trying to determine whether 12-hour bed rest following thrombectomy for ischemic stroke is non-inferior to 24-hour bed rest by measure of outcomes on the modified Rankin Scale (mRS) at 90 days post bed rest.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Received thrombectomy (may have also received intravenous tPA) for a diagnosis of acute ischemic stroke
* TICI 2b/2c/3 score following thromectomy
* Patient and/or Legally Authorized Representative provide consent

Exclusion Criteria:

* TICI 0/1/2a score following thrombectomy
* Venous thromboembolism present at symptom onset
* Pneumonia present at symptom onset
* STEMI at symptom onset
* Positive troponins at symptom onset according to local values
* Bone fracture at symptom onset
* Intubation anticipated or occurred
* Symptomatic intracranial hemorrhage (defined as increase in NIHSS by 4 points or more accompanied by PH2 hemorrhage on imaging) at the time of screening.
* Pre-screening systolic blood pressure < 110 mmHg
* Resting pulse oximetry < 92% (with or without supplemental oxygen)
* Neurological worsening (defined as NIHSS increase of 4 points compared to initial score) prior to screening.
* Baseline modified Rankin Scale score > 2
* Known Pregnancy
* Patient not anticipated to survive 3 months
* Patient not anticipated to follow-up at 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
90 Day Modified Rankin Scale (mRS) score | 90 days post bed rest
  Proportion of patients with a modified Rankin Scale score (min 0, max 5 with 0 being the best outcome) of 0-2 at 90 days

SECONDARY OUTCOMES:
Pneumonia | Duration of hospitalization stay, average 5 days
  Determine whether rates of pneumonia are at least similar in the two arms. Rates will be measured as percentages of the entire population at risk.
Venous Thromboembolism | Duration of hospitalization stay, average 5 days
  Determine whether rates of Venous Thromboembolism (VTE) are at least similar in the two arms. Rates will be measured as percentages of the entire population at risk.
Neurological Worsening | Duration of hospitalization stay, average 5 days
  Determine whether rates of neurological worsening are at least similar in the two arms. Rates will be measured as percentages of the entire population at risk.
Readmission | 90 days post bed rest
  Determine whether rates of readmission are at least similar in the two arms.
Length of Stay | Duration of hospitalization stay, average 5 days
  Determine whether length of hospital stay are at least similar in the two arms. This will be measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Silver, MD, Principal Investigator — UMass Medical School

IPD SHARING:
Plan to Share IPD: No